CLINICAL TRIAL: NCT07022392
Title: Feasibility and Acceptability of the Technology Based Enhanced Gender Support Platform Implementation
Brief Title: Feasibility and Acceptability of the Technology Based Enhanced Gender Support Platform Implementation With Parents
Acronym: TEGS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Gina Sequeira, Assistant Professor, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00005068; K08HS029028-01 (AHRQ)
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Parents; Usability
Keywords: parents

STUDY DESIGN:
Intervention Model Description: All parents and caregivers who agree to participate in the study will receive the same intervention- the TEGS platform. Each will complete surveys at baseline, 1 mo and 3mo after getting access to the platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Technology-Enhanced Gender Support Platform (Experimental)
  Interventions: Other: Technology-enhanced gender support platform

INTERVENTIONS:
Other: Technology-enhanced gender support platform — Technology-based platform to support parents

SUMMARY:
This is a small pilot feasibility and acceptability study of implementing a Technology-Enhanced Gender Support (TEGS) platform with parents and caregivers. Parents and caregivers who consent to participate will complete an electronic survey at baseline. They will then receive access to the TEGS platform and complete follow up surveys 1 mo and 3 mo after. Each participant will also be given the option to participate in an exit interview.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a gender diverse youth aged 8-17
* Has access to the internet
* Can speak or read English

Exclusion Criteria:

* Not a parent of a gender diverse youth aged 8-17
* No access to the internet
* Cannot speak or read in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | 1 month and 3 months
  10 item measure of intervention usability measured on a scale from 0 to 100 with 100 indicating higher usability

SECONDARY OUTCOMES:
Transgender Family Acceptance To Empowerment scale | Baseline, 1 month, 3 month
  16 item measure of parental acceptance and empowerment, measured on a scale of 0 to 80 with 80 indicating a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No